CLINICAL TRIAL: NCT01330602
Title: Intima-Medial Thickness Guidance of Primary Prevention in Relatives of Patients With Early onSet Atherosclerosis: The IMPRESS Study- A Multi-centre, Randomised Controlled Trial
Brief Title: Intima-Medial Thickness Guidance of Primary Prevention in Relatives of Patients With Early onSet Atherosclerosis
Acronym: IMPRESS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: DSRB-C/10/005
Record Dates: First submitted 2010-05-11; First posted 2011-04-07 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Atherosclerotic Cardiovascular Disease; Cardiovascular Disease
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lifestyle counseling (Experimental): All participants randomised into the IMPRESS Intervention group will undergo tailored health profiling.This individual assessment will be carried out within the clinic setting.
  The key elements of the IMPRESS intervention include:
  * Promoting a healthy lifestyle
  * Supporting lifestyle and risk modification
  * Encouraging active self-management of risk and chronic disease
  * Improving coordination of care
  * Pharmacological therapy All the individuals in the intervention group will receive a comprehensive report on their risk status and ideal goals.
  Interventions: Behavioral: IMPRESS intervention
- Usual care arm (No Intervention): Usual Care Following the assessment of absolute cardiovascular risk, usual care participants will be provided a report outlining areas in which improvements could be made for the prevention of atherosclerotic burden.
  No restrictions will be made in respect to usual care management. As such, the prescription of standard medications for primary prevention of atherosclerotic burden based on individual risk factors is anticipated in 20-30% of usual care participants.
  At 18 months and three years those in the usual care arm will be invited to undergo repeat CIMT measurements, pathology, absolute risk score calculation and health-related questionnaires as part of the structured study follow-up

INTERVENTIONS:
Behavioral: IMPRESS intervention — The key elements of the IMPRESS intervention include:
  * Promoting a healthy lifestyle
  * Supporting lifestyle and risk modification
  * Encouraging active self-management of risk and chronic disease
  * Improving coordination of care
  * Pharmacological therapy
  Other Names: Lifestyle medication; CIMT measurement; Statin Therapy; Lifestyle Modification
  Arms: Lifestyle counseling

SUMMARY:
The primary objective of this study is, to instigate a reduction in atherosclerotic burden within the carotid arteries in the intervention group compared to the control group and to demonstrate parallel improvements in cardiovascular and overall health status relative to usual care

DETAILED DESCRIPTION:
Individuals at intermediate risk account for a large proportion of patients presenting with atherosclerotic events. The barriers to reducing this problem relate to the expense of an unselective primary prevention strategy among a group where the majority will not have events, as well as the difficulty of getting apparently well subjects to adhere to lifestyle and pharmacologic management.

An outcome-based study would require large numbers and would be unlikely to be funded without proof of concept. CIMT will be used as a validated surrogate of atherosclerotic status and future cardiovascular events in this study.

As such, this study will use CIMT (as both a delineator of risk and in the primary endpoint), a marker of atherosclerotic burden (the disease process rather than a surrogate), to address the unresolved issue about how to most efficiently manage intermediate risk subjects with a family history of premature atherosclerosis by combining better selection of such individuals for active treatment and recommended lifestyle changes with a DMP strategy to optimise their successful application in the longer-term.

The Intima-Media thickness guidance of Primary prevention in Relatives of individuals with Early onSet atherosclerosiS (IMPRESS) Study will test the following null hypothesis:

In intermediate risk, first-degree relatives (i.e. mother, father, brother or sister) of individuals with premature atherosclerosis, a CIMT-targeted DMP for primary prevention (the IMPRESS intervention) incorporating more intensive non-pharmacological and pharmacological management, provides no better reduction of atherosclerotic burden (as determined by the change in CIMT from baseline to follow-up completion) than usual health care management during three years follow-up.

Study Design The study hypotheses will be examined via a randomised controlled primary prevention/intervention trial comparing an individualised DMP with usual clinical care of middle-aged (40-65 years old) subjects who have a family history of premature cardiovascular disease and are determined to be at intermediate risk for a cardiovascular event within the next 5 years7, 22.

Study Centres

As a multicentre study, participants will be recruited from three centres:

* Princess Alexandra Hospital (Brisbane, Australia): responsible site investigator Associate Professor Karam Kostner
* Baker IDI Heart and Diabetes Institute/ The Alfred Hospital (Melbourne, Australia): responsible site investigator Dr Melinda Carrington
* National University Health System and Novena Heart Centre (Singapore): responsible site investigator Professor Desley Hegney

Participants This study will be conducted in a group of 40-65 year old adults.

IMPRESS Study will test the following null hypothesis:

In intermediate risk, first-degree relatives (i.e. mother, father, brother or sister) of individuals with premature atherosclerosis, a CIMT-targeted DMP for primary prevention (the IMPRESS intervention) incorporating more intensive non-pharmacological and pharmacological management, provides no better reduction of atherosclerotic burden (as determined by the change in CIMT from baseline to follow-up completion) than usual health care management during three years follow-up.

Primary End-Point Consistent with the study hypothesis, the primary study end-point is change in CIMT from baseline to three years, as determined by a blinded core laboratory and analysed on an intention-to-treat basis according to random study group allocation.

Secondary End-Points

The secondary endpoints are change from baseline to three years in the following variables:

i) Plaque length (carotid artery) ii) Internal CIMT iii) General health and well being (as measured by the SF-12 18 and EQ-5D 19) iv) Mental health (as determined by the Arrol 20 +/- CESD 21) v) Health care costs vi) Modifiable risk factors for atherosclerotic disease other than diabetes ( i.e. smoking, dyslipidaemia, obesity and hypertension) vii) Absolute cardiovascular risk profile 22 and risk of diabetes (as determined by the Type 2 Diabetes Risk Assessment Tool [AUSDRISK]) Score 23) viii) Diabetic status (as determined by fasting glucose) ix) All-cause mortality/ cardiovascular hospitalisation

ELIGIBILITY:
Inclusion Criteria:

* Have a first-degree relative (i.e. a mother, father, brother or sister) with premature (onset <65 years of age) atherosclerosis. This includes coronary artery disease/acute myocardial infarction, non-haemorrhagic stroke and peripheral vascular disease.
* Are classified as "intermediate risk" of experiencing a cardiovascular event in the next 5 years as determined via the Framingham Risk Equation 7, 22
* Live within a geographically accessible area for follow-up (i.e. within a 40km radius of the study centre)
* Are living independently in the community or their own home
* Are able and willing to provide written informed consent to participate in the study (this includes the ability to understand and speak English fluently and that the patient is mentally competent)

Exclusion Criteria:

* Pre-existing atherosclerotic disease
* Have been diagnosed with Type 1 or Type 2 Diabetes Mellitus
* Have contraindications to the use of statin medications (includes pregnancy and breastfeeding)
* Unable to provide written informed consent to participate in this study
* Have a terminal malignancy requiring palliative care, or limited life expectancy or any other medical condition (including pregnancy) that results in the belief (deemed by the Chief Investigators) that it is not appropriate for the patient to participate in this trial
* Participating in another clinical research trial

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1310 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change in CIMT from baseline to three years | 3 years
  CIMT will be used as a validated surrogate of atherosclerotic status and future cardiovascular events in this study.
  As such, this study will use CIMT (as both a delineator of risk and in the primary endpoint), a marker of atherosclerotic burden (the disease process rather than a surrogate), to address the unresolved issue about how to most efficiently manage intermediate risk subjects with a family history of premature atherosclerosis

SECONDARY OUTCOMES:
i) Plaque length (carotid artery) ii) Internal CIMT iii) General health and well being iv) Mental health v) Health care costs vi) Modifiable risk factors | 3 years
  In intermediate risk, first-degree relatives (i.e. mother, father, brother or sister) of individuals with premature atherosclerosis, a CIMT-targeted DMP for primary prevention (the IMPRESS intervention) incorporating more intensive non-pharmacological and pharmacological management, provides no better reduction of atherosclerotic burden (as determined by the change in CIMT from baseline to follow-up completion) than usual health care management during three years follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Desley G HEGNEY, Professor, Principal Investigator — National University Health system, NUS
Locations (3):
- Singapore (3):
  - National University Hospital, Singapore
  - Novena heart Centre, Singapore
  - Tan Tock Seng Hospital, Singapore